CLINICAL TRIAL: NCT02087085
Title: Safety and Efficacy of Brimonidine Posterior Segment Drug Delivery System in Patients With Geographic Atrophy Secondary to Age-related Macular Degeneration
Brief Title: A Safety and Efficacy Study of Brimonidine Intravitreal Implant in Geographic Atrophy Secondary to Age-related Macular Degeneration
Acronym: BEACON
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 190342-038; 2013-003320-36 (EudraCT Number)
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-03

CONDITIONS: Geographic Atrophy; Macular Degeneration
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration | interventions — Brimonidine Tartrate; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 400 µg Brimonidine Implant (Experimental): 400 µg brimonidine implant in the study eye, administered by intravitreal injections using the Brimonidine Drug Delivery System (Brimo DDS®) applicator every 3 months from Baseline (Day 1) through Month 21.
  Interventions: Drug: 400 µg Brimonidine Implant
- Sham (Sham Comparator): Sham treatment (control) in the study eye, administered by intravitreal injections using a needleless drug delivery system (DDS) applicator every 3 months from Baseline (Day 1) through Month 21.
  Interventions: Other: Sham

INTERVENTIONS:
Drug: 400 µg Brimonidine Implant — 400 µg brimonidine implant in the study eye using Brimo DDS® applicator on Day 1, and every 3 months through Month 21.
  Other Names: AGN-190342
  Arms: 400 µg Brimonidine Implant
Other: Sham — Sham treatment with needleless applicator (no implant) to the study eye on Day 1, and every 3 months through Month 21.
  Arms: Sham

SUMMARY:
This study will assess the safety and efficacy of the brimonidine intravitreal implant in participants with geographic atrophy due to age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Geographic atrophy due to age-related macular degeneration in the study eye
* Visual acuity better than or equal to 20/125 Snellen equivalent in the study eye and 20/200 Snellen equivalent in the fellow eye.

Exclusion Criteria:

* Cataract surgery or Laser-Assisted in situ Keratomileusis (LASIK) in the study eye in the last 3 months
* Infections in either eye in the last 3 months

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2014-05-09 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Winterson, Study Director — Allergan
Locations (41):
- United States (23):
  - Retinal Consultants of Arizona, Ltd., Retinal Research Institute, Phoenix, Arizona
  - Associated Retina Consultants, Phoenix, Arizona
  - University of California, San Diego, Jacobs Retina Center, Shiley Eye Center, La Jolla, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Retina Consultants of Southern Colorado, PC, Colorado Springs, Colorado
  - "National Ophthalmic Research Institute Retina Consultants of Southwest Florida", Fort Myers, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Southern Vitreoretinal Associates, PL, Tallahassee, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Georgia Retina, Decatur, Georgia
  - Raj K. Maturi, MD, Indianapolis, Indiana
  - Retina Associates of Western New York, Rochester, New York
  - Charlotte Eye Ear Nose & Throat Associates, PA, Charlotte, North Carolina
  - Oregon Retina, LLP, Eugene, Oregon
  - Casey Eye Institute, Oregon Health and Science University, Portland, Oregon
  - Mid Atlantic Retina, Wills Eye Retina Surgeons, Philadelphia, Pennsylvania
  - Retina Research Institute of Texas, Abilene, Texas
  - Texas Retina Associates, Arlington, Texas
  - "Austin Retina Associates ", Austin, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Valley Retina Institute, McAllen, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
- Australia (2):
  - Center for Eye Research Australia, Melbourne, Victoria
  - Lions Eye Institute, University of Western Australia, Nedlands
- France (2):
  - Service d'Ophtalmologie, Bordeaux
  - "Centre Hospitalier Intercommunal de Creteil ", Créteil
- Germany (2):
  - "Universitat Bonn, Abteilung fur Augenheilkunde ", Bonn
  - STZ Eyetrial, Tübingen
- Italy (7):
  - Università di Cagliari (presidio San Giovanni di Dio), Bologna
  - Università di Cagliari (presidio San Giovanni di Dio), Cagliari
  - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - "Dir IV Clinica Oculistica di Milano, Ospedale Generale ""Luigi Sacco"" ", Milan
  - Universita degli Studi di Padova, Dipartimento di Neuroscienze, Padua
  - Universita degli Studi di Torino, Torino
- United Kingdom (5):
  - Clinical Research Unit, Level2, Bristol Eye Hospital, Lower Maudlin Street, Bristol
  - Frimley Park Hospital, Eye clinical trials Unit, Department of Opthalmology, Camberley
  - Moorfields Eye Hospital, London
  - Macular Unit, Hospital of St Cross, Rugby
  - Royal Hallamshire Hospital, Eye Department, Sheffield

REFERENCES:
- [Derived] Miere A, Capuano V, Kessler A, Zambrowski O, Jung C, Colantuono D, Pallone C, Semoun O, Petit E, Souied E. Deep learning-based classification of retinal atrophy using fundus autofluorescence imaging. Comput Biol Med. 2021 Mar;130:104198. doi: 10.1016/j.compbiomed.2020.104198. Epub 2020 Dec 28. PMID 33383315
- [Derived] Kuppermann BD, Patel SS, Boyer DS, Augustin AJ, Freeman WR, Kerr KJ, Guo Q, Schneider S, Lopez FJ; Brimo DDS Gen 1 Study Group. PHASE 2 STUDY OF THE SAFETY AND EFFICACY OF BRIMONIDINE DRUG DELIVERY SYSTEM (BRIMO DDS) GENERATION 1 IN PATIENTS WITH GEOGRAPHIC ATROPHY SECONDARY TO AGE-RELATED MACULAR DEGENERATION. Retina. 2021 Jan 1;41(1):144-155. doi: 10.1097/IAE.0000000000002789. PMID 32134802
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 400 µg Brimonidine Implant | Sham
Started | 154 | 156
Completed | 34 | 40
Not Completed | 120 | 116
Not completed — Adverse Event | 10 | 14
Not completed — Lack of Efficacy | 4 | 3
Not completed — Lost to Follow-up | 6 | 4
Not completed — Withdrawal by Subject | 9 | 11
Not completed — Protocol Violation | 1 | 0
Not completed — Study Terminated by Sponsor | 87 | 80
Not completed — Other Miscellaneous Reasons | 3 | 4

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Sham: Sham treatment (control) in the study eye, administered by intravitreal injections using a needleless DDS applicator every 3 months from Baseline (Day 1) through Month 21.
- Total: Total of all reporting groups
Arm/Group | 400 µg Brimonidine Implant | Sham | Total
Number analyzed (Participants) | 154 | 156 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.9 (7.89) | 77.0 (7.24) | 76.9 (7.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 91 | 192
  Male | 53 | 65 | 118
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 153 | 156 | 309
  Black or African American | 1 | 0 | 1
Geographic Atrophy (GA) Lesion Area by Fundus Autofluorescence (FAF) [Mean (Standard Deviation); unit: millimeters squared (mm^2)] — GA lesion area was measured in mm^2 by FAF and analysis of FAF images was performed by the central reading center. Population: Modified intent-to-treat (mITT) population included all randomized and treated participants with baseline and at least 1 postbaseline assessment for GA lesion area by FAF.
  millimeters squared (mm^2)
    number analyzed (Participants) | 149 | 154 | 303
    (all) | 5.1611 (3.7016) | 5.4761 (3.5961) | 5.3212 (3.6457)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Geographic Atrophy (GA) Lesion Area of the Study Eye as Assessed by Fundus Autofluorescence (FAF) at Month 24
Description: GA lesion area was measured in mm^2 by FAF in the study eye and was quantified by the central reading center. The study eye was defined as the eye that met inclusion/exclusion criteria with the worst standard Best Correct Visual Acuity (BCVA). If the BCVA in both eyes was similar the right eye was selected as the study eye. A positive change from baseline indicates an increase in size of GA lesion area (worsening; disease progression). Mixed model for repeated measures (MMRM) was used for analysis.
Time Frame: Baseline (Day 1) to Month 24
Population: Participants from the mITT population, all randomized and treated participants with baseline and at least 1 postbaseline assessment for GA lesion area by FAF, with data available for analysis at Month 24.
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | 400 µg Brimonidine Implant | Sham
Number analyzed (Participants) | 86 | 90
mm^2 | 3.1455 (0.1377) | 3.5044 (0.1359)
Statistical Analysis 1: Comparison: 400 µg Brimonidine Implant vs Sham; Test type: Superiority; p = 0.047, MMRM — MMRM model included treatment group, study region, analysis visit and treatment-by-visit interaction as factors and baseline value and baseline value-by-analysis visit interaction as covariates; Least Squares Mean Difference = -0.3589, 95% CI 2-sided [-0.7132 to -0.0047], Standard Error of Mean 0.1804

2. Secondary Outcome: Change From Baseline in Standard Best Corrected Visual Acuity (BCVA) Score as Assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) Chart at Month 24
Description: BCVA was measured using an eye chart (ETDRS) and was reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The study eye was defined as the eye that met inclusion/exclusion criteria with the worst standard BCVA. If the BCVA in both eyes was similar the right eye was selected as the study eye. A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening. MMRM was used for analysis.
Time Frame: Baseline (Day 1) to Month 24
Population: Participants from the mITT population, all randomized and treated participants with baseline and at least 1 postbaseline assessment for GA lesion area by FAF, with data available for analysis for this outcome measure at Month 24.
Measure: Least Squares Mean (Standard Error); unit: letters read correctly
Arm/Group | 400 µg Brimonidine Implant | Sham
Number analyzed (Participants) | 81 | 82
letters read correctly | -10.9 (1.0) | -9.7 (1.0)
Statistical Analysis 1: Comparison: 400 µg Brimonidine Implant vs Sham; Test type: Superiority; p = 0.390, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.2, 95% CI 2-sided [-3.9 to 1.5], Standard Error of Mean 1.4

3. Secondary Outcome: Change From Baseline in Low Luminance BCVA Score as Assessed by ETDRS Chart at Month 24
Description: Low Luminance BCVA was measured by placing a 2.0 log unit neutral density filter over the best correction for that eye and having the participant read the normally illuminated ETDRS chart and was reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The study eye was defined as the eye that met inclusion/exclusion criteria with the worst standard BCVA. If the BCVA in both eyes was similar the right eye was selected as the study eye. A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening. MMRM was used for analysis.
Time Frame: Baseline (Day 1) to Month 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: letters read correctly
Arm/Group | 400 µg Brimonidine Implant | Sham
Number analyzed (Participants) | 81 | 82
letters read correctly | -8.1 (1.0) | -6.7 (1.0)
Statistical Analysis 1: Comparison: 400 µg Brimonidine Implant vs Sham; Test type: Superiority; p = 0.301, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -1.4, 95% CI 2-sided [-4.2 to 1.3], Standard Error of Mean 1.4

4. Other Pre Specified Outcome: Change From Baseline in Retinal Sensitivity in the Study Eye
Time Frame: Baseline (Day 1) to Month 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From first dose of study drug to date of last visit (up to approximately 33 months)
Description: Safety population included all participants who received at least 1 administration of study treatment.
Arm/Group | 400 µg Brimonidine Implant | Sham
All-Cause Mortality (participants affected / at risk) | 5/154 | 6/156
Serious Adverse Events (participants affected / at risk) | 48/154 | 37/156
Other Adverse Events (participants affected / at risk) | 79/154 | 61/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 400 µg Brimonidine Implant (N=154) | Sham (N=156)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 1
Bradycardia (Cardiac disorders) | 3 | 0
Cardiac failure congestive (Cardiac disorders) | 3 | 1
Coronary artery disease (Cardiac disorders) | 2 | 1
Sinus node dysfunction (Cardiac disorders) | 2 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 2 | 0
Vitreous haemorrhage (Eye disorders) | 2 | 0
Retinal tear (Eye disorders) | 1 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0
Anterior capsule contraction (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Spigelian hernia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Hernia (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 3
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 2
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Flail chest (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Acquired claw toe (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Desmoplastic melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain stem ischaemia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dementia alzheimer's type (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Device dislocation (Product Issues) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 2
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 400 µg Brimonidine Implant (N=154) | Sham (N=156)
Vitreous floaters (Eye disorders) | 29 | 1
Conjunctival haemorrhage (Eye disorders) | 21 | 11
Visual impairment (Eye disorders) | 12 | 6
Eye pain (Eye disorders) | 11 | 9
Visual acuity reduced (Eye disorders) | 9 | 6
Dry eye (Eye disorders) | 8 | 6
Ocular discomfort (Eye disorders) | 8 | 1
Nasopharyngitis (Infections and infestations) | 12 | 12
Urinary tract infection (Infections and infestations) | 3 | 15
Fall (Injury, poisoning and procedural complications) | 5 | 10
Headache (Nervous system disorders) | 8 | 4
Hypertension (Vascular disorders) | 8 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT02087085/SAP_000.pdf
  • Study Protocol (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT02087085/Prot_001.pdf